CLINICAL TRIAL: NCT00030147
Title: The Efficacy of Phytoestrogens and Selective Estrogen Receptor Modulators in Perimenopause-Related Depression
Brief Title: Raloxifene and Rimostil for Perimenopause-Related Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 020120; ZIAMH002537-26 (NIH); 02-M-0120 (Other: NIHCC)
Record Dates: First submitted 2002-02-06; First posted 2002-02-07 (Estimated); Results first posted 2016-09-05 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-07

CONDITIONS: Perimenopausal Depression; Depression
Keywords: Gonadal Steroids; Estrogen Receptor; Mood Disorders; Perimenopause; Estradiol; Depression; Estrogen Response Element; Perimenopausal; Perimenopausal Depression
MeSH Terms: conditions — Depression; Mood Disorders | interventions — Raloxifene Hydrochloride; Estradiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Raloxifene (Experimental): Raloxifene (Evista) 60 mg per day and placebo skin patch for eight weeks
  Interventions: Drug: Raloxifene
- Rimostil (Experimental): Rimostil (phytoestrogen) 1000 mg twice a day and placebo skin patch for eight weeks
  Interventions: Drug: Rimostil
- Transdermal estradiol (Active Comparator): 17-beta estradiol 100 micrograms a day by skin patch and placebo tablets for eight weeks
  Interventions: Drug: Transdermal Estradiol
- Placebo (Placebo Comparator): Placebo skin patch and placebo tablets for eight weeks.
  Interventions: Drug: Placebo skin patch and placebo tablets

INTERVENTIONS:
Drug: Raloxifene — 60 mg a day orally administered
  Other Names: Evista
  Arms: Raloxifene
Drug: Rimostil — 1000 mg twice a day administered orally
  Arms: Rimostil
Drug: Transdermal Estradiol — 100 microgram per day transdermal estradiol
  Other Names: Alora
  Arms: Transdermal estradiol
Drug: Placebo skin patch and placebo tablets — matched placebo skin patch to transdermal estradiol and matched tablets to either Raloxifene or Rimostil
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the drugs raloxifene and rimostil in treating perimenopause-related depression.

Perimenopause-related mood disorders cause significant distress to a large number of women; the demand for effective therapies to treat these mood disorders is considerable. Estradiol replacement therapy (ERT) has demonstrated efficacy in treating perimenopause-related depression. Unfortunately, there are long-term risks associated with ERT. Selective estrogen receptor modulators (SERMS), such as raloxifene, and phytoestrogens, such as rimostil, have estrogen-like properties and may offer a safer alternative to ERT. The effect of SERMS and phytoestrogens on mood and cognitive functioning need to be examined in women with perimenopause-related depression.

Participants in this study will undergo a medical history, physical examination, electrocardiogram (EKG), and blood and urine tests. They will then be randomly assigned to receive one of four treatments for 8 weeks: raloxifene pills plus a placebo (an inactive substance) skin patch, rimostil pills plus placebo skin patch, estradiol skin patch plus placebo pills, or placebo patch plus placebo pills. Participants will have clinic visits every 2 weeks. During the visits, blood will be drawn and participants will meet with staff members and complete symptom self-rating scales. A urine and blood sample will be collected at the beginning and end of the study. At the end of the study, participants who received placebo or whose study medication was ineffective will be offered treatment with standard antidepressant medications for 8 weeks. Non-menstruating women will receive progesterone for 10 days to induce menstrual bleeding and shedding of the inner layer of the uterus, which may have been stimulated by the study medications.

DETAILED DESCRIPTION:
Perimenopause-related mood disorders cause significant distress to a potentially large number of women. The demand for effective therapeutic alternatives to estrogen for treating these mood disorders is considerable, as is the need to define clinical or biologic markers that may predict successful response of mood disturbances to phytoestrogens or selective estrogen receptor modulators (SERMs). Further, the study of potential biological mechanisms underlying both perimenopause-related mood disorders and their response to treatment may offer the possibility of uncovering some etiopathogenic mechanisms involved in these and related mood disorders.

Results of protocol # 90-M-0077 demonstrated the therapeutic efficacy of estradiol therapy (ET) in perimenopausal depression, independent of its effects on vasomotor symptoms. Nevertheless, the long term risks of ET to endometrial and breast tissues continue to deter many women from its use. Recently, selective estrogen receptor modulators (SERMs) and phytoestrogens (plant-derived estrogen-like compounds) have become available and are reported to display both tissue-specific profiles of estrogen agonist and antagonist actions and differential affinities for the two forms of estrogen receptor. For many women, these novel compounds would represent a safer alternative to ET for the prevention of osteoporosis and the treatment of menopausal symptoms. However, the effects of SERMs and phytoestrogens on mood and cognitive function in perimenopausal women remain undetermined.

In this protocol we wish both to investigate the effects of SERMs and phytoestrogens on mood and cognition under placebo controlled conditions and to compare these effects with estradiol therapy. This protocol will address the following questions: 1) Do selective estrogen receptor modulators or phytoestrogens improve mood and cognition in perimenopausal depressed women? 2) Are the mood and cognitive effects of SERMs and phytoestrogens comparable to those of ET? and 3) Do selective estrogen receptor modulators and phytoestrogens improve measures of bone metabolism in perimenopausal depressed women?

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects for this study will meet the following criteria:

1. Self-report of the onset of depression associated with menstrual cycle irregularity or amenorrhea;
2. A current episode of minor (meeting 3-4 criterion symptoms) or major depression (of moderate severity or less on the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV (SCID) severity scale and not meeting DSM-IV criteria symptom 9 (suicide)) as determined by the administration of the minor depression module of the Schedule for Affective Disorders and Schizophrenia - Lifetime Version (SADS-L). Additionally, to ensure that subjects meet a minimum threshold for severity of depression, subjects will have scores greater than or equal to 10 on either the Beck Depression Inventory (BDI) or the Center for Epidemiologic Studies - Depression (CES-D) Scale during at least three of the four clinic visits during the two month screening phase, as well as a 17 item Hamilton Depression score greater than or equal to 10. Subjects will be excluded if they meet any of the following criteria: major depression of greater than moderate severity, DSM-IV criteria # 9 (suicide), or anyone requiring immediate treatment after clinical assessment or functional impairment ratings of five or six for more than seven consecutive days on daily ratings;
3. Evidence of perimenopausal reproductive status;
4. Age 40 to 60;
5. No prior hormonal therapy for the treatment of perimenopause-related mood or physical symptoms within the last six months;
6. No history of psychiatric illness during the two years prior to the reported onset of the current episode of depression;
7. In good medical health, and not taking any medication or dietary and herbal supplements on a regular basis (with the exception of multivitamins and calcium supplements).

EXCLUSION CRITERIA:

The following conditions will constitute contraindications to treatment and will preclude a subject s participation in this protocol:

1) Severe major depression with any of the following:

1. positive (threshold) response to SCID major depression section item # 9, suicidal ideation;
2. anyone requiring immediate treatment after clinical assessment;
3. severity ratings greater than moderate on the SCID IV interview;
4. functional impairment ratings of five or six for more than seven consecutive days on daily ratings.

2) Current treatment with antidepressant medications. Our main concern is to exclude subjects taking medications that would treat or precipitate depression or adversely interact with reproductive hormones, phytoestrogens (e.g., anticoagulants), or SERMs. Thus, we wish to exclude only women receiving psychotropic medications, medications that have been reported to induce a change in mood or behavior, hormone replacement therapy, oral contraceptive agents, or medications that may have a potential adverse interaction with the compounds employed in this study.

3) History of psychiatric illness during the two years before the reported onset of the current episode of depression.

4) History of ischemic cardiac disease, pulmonary embolism, retinal thrombosis, or thrombophlebitis; any subject with risk factors for thrombo-embolic phenomena including cigarette smokers; varicose veins, patients with prolonged periods of immobilization (including prolonged travel), and active heart disease. The literature suggests that although both smoking and hormone replacement/oral contraceptives have associated risks of thromboembolic phenomena and cardiovascular events, these individual risks do not become significantly greater when combined until greater than 10 cigarettes a day are consumed. Thus we wish to exclude only subjects for this study who smoke greater than 10 cigarettes per day.

5) Renal disease, asthma.

6) Hepatic dysfunction.

7) Women with a history of carcinoma of the breast, or any women with a family history of the following: premenopausal breast cancer or bilateral breast cancer in a first degree relative; multiple family members (greater than three relatives) with postmenopausal breast cancer.

8) Women with a history of uterine cancer, endometriosis, ill-defined pelvic lesions, particularly undiagnosed ovarian enlargement, undiagnosed vaginal bleeding.

9) Patients with a known hypersensitivity to raloxifene, phytoestrogens (including Rimostil, isoflavones, genistein, daidzein, red clover extract and soy-related compounds), estradiol, Alora, medroxyprogesterone acetate, or the excipients (inactive compounds) contained within these medications including: Rimostil -tocopherols, cellulose, calcium hydrogen phosphate, magnesium stearate, silica-colloidal anhydrous; Provera - calcium stearate, corn starch, lactose, mineral oil, sorbic acid, sucrose, talc; Alora - sorbitan monooleate, acrylic adhesive; Evista - anhydrous lactose, carnauba wax, crospovidone, Federal Food, Drug, and Cosmetic Act (FD& C) blue # 2 aluminum lake, hydroxypropyl methylcellulose, lactose monohydrate, magnesium stearate, modified pharmaceutical glaze, polyethylene glycol, polysorbate 80, povidone, and titanium dioxide.

10) Pregnant women.

11) Porphyria.

12) Diabetes mellitus.

13) Cholecystitis or pancreatitis.

14) History of cerebrovascular disease (stroke), epilepsy, hypertension, hypercalcemia.

15) Recurrent migraine headaches.

16) Malignant melanoma.

17) History of familial hyperlipoproteinemia.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2002-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Schmidt, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schmidt PJ, Wei SM, Martinez PE, Dor RRB, Guerrieri GM, Palladino PP, Harsh VL, Li HJ, Wakim P, Nieman LK, Rubinow DR. The short-term effects of estradiol, raloxifene, and a phytoestrogen in women with perimenopausal depression. Menopause. 2021 Jan 15;28(4):369-383. doi: 10.1097/GME.0000000000001724. PMID 33470755
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2002-M-0120.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants signed the consent but were not started (did not meet inclusion criteria.)
Groups:
- Estradiol: Transdermal estradiol 17-beta estradiol 100 micrograms a day by skin patch and placebo tablets for eight weeks
- Rimostil: Rimostil (phytoestrogen) 1000mg twice a day and placebo skin patch for eight weeks
Period: Overall Study
Arm/Group | Estradiol | Placebo | Raloxifene | Rimostil
Started | 17 | 19 | 16 | 11
Completed | 17 | 18 | 16 | 11
Not Completed | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Estradiol | Placebo | Raloxifene | Rimostil | Total
Number analyzed (Participants) | 17 | 19 | 16 | 11 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 19 | 16 | 11 | 63
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 16 | 11 | 63
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 2 | 0 | 6
  Not Hispanic or Latino | 15 | 16 | 14 | 10 | 55
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 7 | 1 | 0 | 12
  White | 13 | 9 | 13 | 9 | 44
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Center for Epidemiologic Studies-Depression Scale (CES-D)
Description: Center for Epidemiologic Studies-Depression Scale (CES-D) cutoff scores are typically used as a screen to identify clinically significant depression; a cutoff score of greater than 16 has been shown to correlate with clinically significant depression. In addition, a score between 8 and 15 has been used to define subsyndromal depression. The possible range of scores is zero to 60, with the higher scores indicating more symptoms, weighted by frequency of occurrence during the past week.
Time Frame: Baseline
Population: The analyses included those subjects who started the study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Estradiol | Placebo | Raloxifene | Rimostil
Number analyzed (Participants) | 17 | 19 | 16 | 11
Units on a scale | 27.4 (5.76) | 29.1 (9) | 28.8 (7.9) | 24.6 (5.5)

2. Primary Outcome: Center for Epidemiologic Studies-Depression Scale (CES-D)
Description: as for outcome 1
Time Frame: Week 8
Population: The analyses included those subjects who completed eight weeks of study
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Estradiol | Placebo | Raloxifene | Rimostil
Number analyzed (Participants) | 16 | 17 | 16 | 11
Units on a scale | 9.6 (9.4) | 10.5 (11.3) | 15.8 (8.9) | 16.1 (8.8)

ADVERSE EVENTS:
Arm/Group | Estradiol | Placebo | Raloxifene | Rimostil
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/19 | 0/16 | 0/11
Other Adverse Events (participants affected / at risk) | 1/17 | 2/19 | 1/16 | 0/11
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Estradiol (N=17) | Placebo (N=19) | Raloxifene (N=16) | Rimostil (N=11)
Allergic reaction (Immune system disorders) | 0 | 1 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Two participants signed the consent but were not started (did not meet inclusion criteria.) Early termination of Rimostil treatment arm limits the generalizability of treatment response in this arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes